CLINICAL TRIAL: NCT04041908
Title: Observation of the Use of a Medical Food in Older Adults Undergoing Surgery
Brief Title: Use of a Medical Food in Adults Undergoing Surgery
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low enrollment
Sponsor: Abbott Nutrition (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: BL42
Record Dates: First submitted 2019-07-30; First posted 2019-08-01 (Actual); Last update posted 2020-05-01 (Actual); Status verified 2020-04

CONDITIONS: Compliance, Patient
MeSH Terms: conditions — Patient Compliance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental Product (Experimental): Drink mix powder
  Interventions: Other: Experimental Product

INTERVENTIONS:
Other: Experimental Product — 2 sachets per day

SUMMARY:
Multi-center, prospective, one arm study to evaluate the addition of a medical food to the standard of care in elderly adults undergoing a surgical procedure.

ELIGIBILITY:
Inclusion Criteria:

* Participant is scheduled to have non-melanoma skin cancer on either the head, leg, trunk and arm removed with final wound size of 1.0 to < 5.0 cm in diameter or with 1.0 < 5.0 cm long axis if not circular that will be healed by secondary intent
* Participant has an acceptable state of health and nutrition
* Participant agrees not to begin taking any new medications, dietary supplements, or alternative therapies during the study period
* Participant is interested in participating in the study, willing to comply with the study protocol, and willing to consume two servings of drink mix per day according to the protocol
* Participant has voluntarily signed and dated an informed consent form (ICF), approved by an Independent Ethics Committee/Institutional Review Board (IEC/IRB) and provided Health Insurance Portability and Accountability (HIPAA) authorization prior to any study participation

Exclusion Criteria:

* Participant has a disease or condition that could interfere with the assessment of safety and efficacy of the study treatment and compliance of the participant with study visits/procedures
* Participant has type 1 diabetes mellitus or uncontrolled type 2 diabetes mellitus
* Participant has known immunosuppression
* Participant has platelet or coagulation disorders
* Therapy with another investigational agent within 30 days of Visit 1 that has not been approved
* Systemic infection at the time of enrollment in the study
* Currently receiving or have received recombinant human platelet-derived growth factor or similar therapies, or other bioengineered tissue therapy within the previous 4 weeks
* Participant has an allergy or intolerance to any ingredient in the study product
* Participant is taking nutritional supplement(s)/capsules/formulas for wound healing and is unwilling to discontinue therapy for the duration of the study
* Participation in another clinical study

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2020-03-13 (Actual); Primary Completion 2020-04-10 (Actual); Study Completion 2020-04-10 (Actual)

PRIMARY OUTCOMES:
Product Compliance | Study Day 1 to Study Day 30
  Percent of required study product intake from subject completed intake questionnaire

SECONDARY OUTCOMES:
Investigator Wound Assessment | Study Day 1 to Study Day 30
  Percent of patients with complete wound healing based on physician assessment
Participant Wound Assessment Questionnaire | Study Day 14 and Study Day 30
  Participant completed 4 questions related to wound healing experience; 3 Likert-type questions scaled from 1-10 in negative direction; 1 dichotomous scale question

OTHER OUTCOMES:
Product Evaluation Questionnaire | Study Day 30/Exit
  Participant completed questionnaire; 4 Likert-type questions scaled from 1 - 9 in the negative direction; 2 Likert-type questions scaled from 1 - 5 in the negative direction

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Nelson, PhD, Study Chair — Abbott Nutrition
Locations (1):
- ClinOhio Research Services, Columbus, Ohio, United States